CLINICAL TRIAL: NCT02814500
Title: DP-R212 Pharmacokinetic Study Pharmacokinetic Characteristics of DP-R212 in Comparison to Each Component Coadministered in Healthy Volunteers
Brief Title: DP-R212 Pharmacokinetic Study Phase I
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR-212-I-02
Record Dates: First submitted 2016-06-12; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A group (Experimental): Amlodipine and Rosuvastatin, DP-R212
  Interventions: Drug: DP-R212; Drug: Amlodipine; Drug: Rosuvastatin
- B group (Experimental): DP-R212, Amlodipine and Rosuvastatin
  Interventions: Drug: DP-R212; Drug: Amlodipine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: DP-R212 — Investigational product is prescribed to all of randomized subjects
Drug: Amlodipine — Investigational product is prescribed to all of randomized subjects
Drug: Rosuvastatin — Investigational product is prescribed to all of randomized subjects

SUMMARY:
An open label, randomized, 2-sequence, 2-period, single-dose cross-over study to evaluate the pharmacokinetics characteristics of DP-R212

DETAILED DESCRIPTION:
An open label, randomized, 2-sequence, 2-period, single-dose cross-over study to evaluate the pharmacokinetics characteristics of DP-R212, a fixed dose combination compared with coadministration of separate constituents in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* BMI 17.5~30.5
* signed the informed consent form prior to the study participation

Exclusion Criteria:

* Clinically significant disease
* Previously donate whole blood within 60 days or component blood within 30 days
* Clinically significant allergic disease
* Taken IP in other trial within 90 days
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
AUClast | 0,0.5,1, 2, 3, 4, 5, 6, 8, 10, 12, 24,48,72 hr
Cmax | 0,0.5,1, 2, 3, 4, 5, 6, 8, 10, 12, 24,48,72 hr

IPD SHARING:
Plan to Share IPD: Undecided